CLINICAL TRIAL: NCT04752228
Title: Adverse Childhood Experiences in Patients With Coronary Artery Disease: a Pilot Randomized Control Trial
Brief Title: Adverse Childhood Experiences in Patients With Coronary Artery Disease Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Socar Research SA (Network)
Responsible Party: Principal Investigator, Michael Farkouh, Vice-Chair Research & Professor of Medicine, Department of Medicine, University of Toronto, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-5967
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Adverse Childhood Experiences; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACE Screen (Experimental): At the initial visit, the Philadelphia ACE Survey, a validated ACE questionnaire, will be administered by a research coordinator. A Lifestyle Assessment package will also be provided for self-completion, featuring General Demographics, Cardiovascular and Medication History, Health Behaviours, the Short Form (36) Health Survey, the Patient Health Questionnaire-9, the General Anxiety Disorder-7 questionnaire, the Seattle Angina Questionnaire-7, and the modified Perceived Need for Card Questionnaire. Patients who test positive for ACE will receive a 3-page printed ACE Resource Pack.
  At 3 months, the Lifestyle Assessment will be administered again.
  At 6 months, the Philadelphia ACE survey, Lifestyle Assessment, as well as a scale assessing their comfort level in being screened for ACE, disclosing their ACE status to their clinicians, and their confidence level in their clinicians' ability to help them manage their ACEs will be administered.
  Interventions: Other: Philadelphia ACE Survey; Other: Lifestyle Assessment
- Lifestyle Assessment (Other): At the initial visit, no Philadelphia ACE Survey will be administered. The Lifestyle Assessment packaged will be provided for self-completion, featuring General Demographics, Cardiovascular and Medication History, Health Behaviours, the Short Form (36) Health Survey, the Patient Health Questionnaire-9, the General Anxiety Disorder-7 questionnaire, the Seattle Angina Questionnaire-7, and the modified Perceived Need for Card Questionnaire.
  At 3 months, the Lifestyle Assessment will be administered again.
  At 6 months, the Philadelphia ACE survey, Lifestyle Assessment, as well as a scale assessing their comfort level in being screened for ACE, disclosing their ACE status to their clinicians, and their confidence level in their clinicians' ability to help them manage their ACEs will be administered.
  Interventions: Other: Lifestyle Assessment

INTERVENTIONS:
Other: Philadelphia ACE Survey — The Philadelphia ACE survey assesses the three major domains featured within the original ACE Study Questionnaire developed by Felitti et al. (abuse, neglect, and family dysfunction), in addition to five community-level stressors.
  Arms: ACE Screen
Other: Lifestyle Assessment — The Lifestyle Assessment questionnaire features the Short Form (36) Health Survey, Patient Health Questionnaire-9, General Anxiety Disorder-7 questionnaire, Seattle Angina Questionnaire-7, and modified Perceived Need for Card Questionnaire, which are validated questionnaires for the assessment of quality of life, depression, anxiety, angina, and perceived need for care, respectively.

SUMMARY:
Adverse Childhood Experiences (ACEs) are potentially harmful events occurring during childhood that have been associated with chronic physical conditions in adulthood, including coronary artery disease (CAD). ACEs may constitute a portion of the remaining unexplained residual risk for CAD in adults. Identifying a means of addressing these experiences may mitigate their health consequences and result in improved cardiovascular outcomes.

The primary objective of this study is to determine if patients who undergo ACE screening experience improved quality of life compared to patients who undergo conventional lifestyle assessment.

This will be a single-centre, pragmatic, single-blinded (i.e. data analysts), 1:1, pilot randomized control trial.

DETAILED DESCRIPTION:
ACEs encapsulate a broad spectrum of traumatic and distressing events occurring before the age of 18 that span the domains of abuse, household dysfunction, neglect, amongst others, and that threaten a child's physical, familial or social safety. The landmark ACE Study, published by Felitti and colleagues, was the first study to propose the association between ACEs and the development of chronic physical conditions in adulthood, including cardiovascular disease (CVD). Due to a variety of mechanisms, exposure to an ACE increases predisposition to the development of CVD and its conventional risk factors. ACEs nonetheless remain underrecognized and undermanaged in routine cardiovascular clinical encounters.

Integration of ACE screening into the standardized clinical assessment of CVD may enable cardiologists to better identify patients who might benefit from further post-ACE resiliency interventions and serve as an impactful secondary and tertiary prevention strategy. The ACE screening process itself may be therapeutic as it gives patients the opportunity to discuss their early experiences, reflect on the role of early adversity in their current health problems, and have some sympathetic acknowledgement about this history from a health care professional. This has been termed "ACE insight". Screening for ACEs has been found to be acceptable by patients. Patients may have never had any opportunity to discuss ACEs they have undergone throughout their entire life, enabling their effects to propagate into adulthood. Inquiring about ACE exposure during clinical encounters with all patients may garner insights that can have a beneficial effect in improving cardiovascular health. Additionally, engaging patients in stress-coping therapies, such as mindfulness, and referral for psychological consultation as needed, may also be helpful. Although logical, these strategies still lack adequate evidence and a randomized trial is needed to evaluate their potential in reducing the occurrence of cardiovascular events.

This study aims to assess whether deleterious childhood exposures are associated with an increased prevalence of risk factors for CAD and represent an independent risk factor for CAD. Furthermore, screening for ACEs in patients with CAD may serve as a therapeutic intervention in itself by providing both ACE insight and a platform to unload internal psychological burdens. Screening may result in an enhanced quality of life, as well as improved health behaviours that may benefit their cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at screening
2. History of (1) acute coronary syndrome (ACS) OR (2) coronary artery disease (CAD) necessitating prior cardiovascular intervention. History of ACS determined by documentation of ST-elevation myocardial infarction or non-ST-segment elevation infarction 1-12 months prior to time of screening. History of CAD determined by documentation of percutaneous coronary intervention or coronary artery bypass surgery within the last 1-12 months.
3. Able to complete a survey independently
4. Access to a phone
5. Willingness to participate as evidenced by signing of the study informed consent form

Exclusion Criteria:

1. Inability to speak, read and write in English
2. Cognitive impairment
3. Severe physical or mental illness
4. Limited life expectancy (projected to be less than 1 year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Patient-reported quality of life | 3 and 6 months
  Degree of change in quality of life measured by the Short Form (36) Health Survey questionnaire

SECONDARY OUTCOMES:
Mortality | 6 months
  Rate of all-cause mortality
Cardiovascular hospitalization | 6 months
  Rate of hospitalization for ACS, heart failure, stroke and atrial fibrillation
Myocardial infarction | 6 months
  Rate of myocardial infarction
Stroke | 6 months
  Rate of stroke
Need for urgent repeat coronary revascularization | 6 months
  Rate of need for urgent repeat coronary revascularization

OTHER OUTCOMES:
Health behaviour | 3 and 6 months
  Change in health behaviours, measured using constructs derived from the American Heart Association
Depression | 3 and 6 months
  Change in severity of depression, measured using the Patient Health Questionnaire 9
Anxiety | 3 and 6 months
  Change in severity of anxiety, measured using the Generalized Anxiety Disorder-7 scale
Angina | 3 and 6 months
  Change in angina, measured by the Seattle Angina Questionnaire
Perceived need for care | 3 and 6 months
  Change in perceived need for care, measured by the Modified Perceived Need for Care Questionnaire
Prevalence of ACE | 0 and 6 months
  Percentage of patients with CAD who report history of ACE
Patient preferences on ACE screening | 6 months
  Scale assessing comfort level in being screened for ACE, disclosing their ACE status to their clinicians, and their confidence level in their clinicians' ability to help them manage their ACEs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farkouh, MD, Principal Investigator — University Health Network-Toronto General Hospital, Canada; Claudia Frankfurter, MD, Principal Investigator — University Health Network-Toronto General Hospital, Canada; Lucas C Godoy, MD, Principal Investigator — University Health Network-Toronto General Hospital, Canada; Christine Lay, MD, Principal Investigator — Women's College Hospital, Canada; Robert Maunder, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Peter Munk Cardiac Centre - University Health Network, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Godoy LC, Frankfurter C, Cooper M, Lay C, Maunder R, Farkouh ME. Association of Adverse Childhood Experiences With Cardiovascular Disease Later in Life: A Review. JAMA Cardiol. 2021 Feb 1;6(2):228-235. doi: 10.1001/jamacardio.2020.6050. PMID 33263716
- [Background] Maunder RG, Hunter JJ, Tannenbaum DW, Le TL, Lay C. Physicians' knowledge and practices regarding screening adult patients for adverse childhood experiences: a survey. BMC Health Serv Res. 2020 Apr 15;20(1):314. doi: 10.1186/s12913-020-05124-6. PMID 32293444
- [Background] Maunder RG, Tannenbaum DW, Permaul JA, Nutik M, Haber C, Mitri M, Costantini D, Hunter JJ. The prevalence and clinical correlates of adverse childhood experiences in a cross-sectional study of primary care patients with cardiometabolic disease or risk factors. BMC Cardiovasc Disord. 2019 Dec 19;19(1):304. doi: 10.1186/s12872-019-01277-3. PMID 31881981